CLINICAL TRIAL: NCT07050251
Title: Bridging the Divide: A Pioneering Culturally-Specific Mentoring Intervention to Increase Support for At-Risk Youth
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Jarrad Hodge, Postdoctoral Research Fellow, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-24-1243
Record Dates: First submitted 2025-06-25; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Socio-emotional Well-being; Psychological Well-Being
Keywords: at risk youth; Boys and Girls Clubs
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mentoring Intervention Delivery (Experimental)
  Interventions: Behavioral: Mentoring Intervention Delivery

INTERVENTIONS:
Behavioral: Mentoring Intervention Delivery — The intervention will utilize a culturally specific, socio-emotional learning (SEL) curriculum, adapted based on feedback from the focus groups. The intervention will consist of 10 weekly mentoring sessions lasting 1 hour each. Licensed clinicians will lead sessions and will also serve as mentors.

SUMMARY:
The purpose of this study is to assess the feasibility, acceptability, and effectiveness of a culturally-specific mentoring intervention to improve socio-emotional skills, psychological well-being, and social support among at-risk youth and to evaluate the proposed mentoring intervention's impact on academic outcomes, social behavior, and caregiver perceptions of social-emotional competencies. Additionally, it seeks to gather stakeholder feedback to refine the intervention further.

ELIGIBILITY:
Inclusion Criteria:

* actively enrolled in the partnering community organization (e.g., Boys and Girls Clubs)
* Participants and their caregivers must be able to provide informed assent/consent in English. Parental Consent: Participants must have parental or guardian consent to participate in the study.
* Self-identifies as a racial-ethnic minority (i.e., Black/African American, Hispanic, etc.)

Exclusion Criteria:

* Current participation in another mentoring program: To avoid confounding the results, youth currently involved in other mentoring or structured socio-emotional support programs will be excluded.
* Severe cognitive or developmental disabilities: The study will exclude participants with mental impairments that prevent meaningful engagement in focus groups or intervention activities.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-06-27 (Estimated); Primary Completion 2025-07-26 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Change in Social Emotional Competence as measured by the Social Emotional Competence Questionnaire (SECQ) | Baseline, post-intervention (at 10 weeks)
  The SECQ consists of 25 items, divided into five domains:Self-Awareness, Social Awareness, Self-Management, Relationship Skills and Responsible Decision-Making.Each domain includes 5 items and each is scored from 1(never) to 5 (always) for a maximum score of 25 for each domain. An average of all 25 item responses is calculated and score range is 1.0-5.0, higher score indicating greater social emotional competence.
Change in Parenting Sense of Competence as measured by the Parenting Sense of Competence Scale (PSOC) | Baseline, post-intervention (at 10 weeks)
  The Parenting Sense of Competence Scale (PSOC) contains 16 items and each is scored on a 6-point Likert scale from 1 (Strongly Disagree) to 6 (Strongly Agree) for a maximum score of 96, higher scores indicating greater parenting competence.
Change in Psychological Well-Being as measured by Psychological Well-Being (Ryff's 18-item) assessment | Baseline, post-intervention (at 10 weeks)
  Ryff's 18-item Psychological Well-Being Scale assesses six dimensions of well-being: autonomy, environmental mastery, personal growth, positive relations with others, purpose in life, and self-acceptance. Each subscale consists of 3 items, rated on a 6-point Likert scale from "Strongly Disagree" (1) to "Strongly Agree" (6). Maximum score is 108 and higher scores indicate greater psychological well-being.
Change in depression, anxiety, and stress symptoms as measured by the Depression Anxiety Stress Scale (DASS-21) | Baseline, post-intervention (at 10 weeks)
  DASS-21) is a validated self-report questionnaire that assesses symptoms across three domains: depression, anxiety, and stress. Each domain consists of 7 items rated on a 4-point Likert scale from 0 (Did not apply to me at all)-3( Applied to me very much, or most of the time). Scores for each domain are summed and then multiplied by 2 to match the original DASS-42 scale for a maximum score of 126. Higher scores indicate greater symptom severity.

SECONDARY OUTCOMES:
Change in Academic Self-Efficacy as measured by the Academic Self-Efficacy Scale (ASES) | Baseline, post-intervention (at 10 weeks)
  ASES consists of 9 items, each rated on a 5-point Likert scale from 1(not at all confident) to 5(extremely confident) for a maximum score of 45. Higher scores indicate greater academic self-efficacy
Change in emotional and behavioral functioning as measured by the Strengths and Difficulties Questionnaire (SDQ) | pre- and post-intervention assessments (at 10 weeks).
  SDQ consists of 25 items across five subscales: emotional symptoms, conduct problems, hyperactivity/inattention, peer relationship problems, and prosocial behavior. Each item is rated on a 3-point scale from 0 (Not True), 1 (Somewhat True) , 2 (Certainly True) for a maximums score of 40 for the Emotional Symptoms, Conduct Problems, Hyperactivity/Inattention, and Peer Relationship Problems subscales and higher score indicates greater difficulties. the Prosocial Behavior subscale has a score range from 0-10 and higher score indicate more positive social behavior.
Change in perceived social support as measured by the Multidimensional Scale of Perceived Social Support (MSPSS) | pre- and post-intervention assessments (at 10 weeks).
  MSPSS consists of 12 items, with 4 items in each domain, rated on a 7-point Likert scale from 1 (Very Strongly Disagree) to 7 (Very Strongly Agree) for a maximum of score of 84. Higher scores indicate greater perceived social support.
Change in well-being as measured by the Multidimensional Well-Being Assessment (MWBA) | pre- and post-intervention assessments (at 10 weeks).
  This is a 30 item questionnaire with each item scored from 1( not at all) to 5 (very often), for a maximum total score of 150. Higher scores indicate better well-being.

CONTACTS AND LOCATIONS:
Overall Officials: Jarrad Hodge, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No